CLINICAL TRIAL: NCT04813055
Title: Prospective Registry Of Therapeutic EndoscopiC ulTrasound
Acronym: PROTECT
Status: Recruiting | Type: Observational
Sponsor: Paolo Giorgio Arcidiacono, MD (Other)
Responsible Party: Sponsor-Investigator, Paolo Giorgio Arcidiacono, MD, Prof. Dr., IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: 178/INT/2020
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastric Outlet Obstruction; Biliary Obstruction; Acute Pancreatic Fluid Collection; Acute Pancreatitis With Infected Necrosis; Acute Cholecystitis; Chronic Pancreatitis
Keywords: Endoscopic ultrasound; Therapeutic EUS; Interventional EUS; Biliary Drainage; Gastro-jejunostomy; Gallbladder Drainage; Endoscopy
MeSH Terms: conditions — Gastric Outlet Obstruction; Cholecystitis, Acute; Pancreatitis, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapeutic EUS: Procedures involving Linear Echoendoscopes to create a communication between the gastrointestinal tract and a target organ (biliary tree, pancreatic duct, fluid collection, gallbladder, downstream gastrointestinal tract) through plastic or metal stents.
  Interventions: Procedure: Therapeutic EUS
- Controls: Patients eligible for T-EUS procedures, but undergoing alternative surgical interventions, percutaneous interventions (e.g. Percutaneous Biliary Drainage) or non-EUS based endoscopic procedures (e.g. enteral stenting)
  Interventions: Procedure: Percutaneous Procedures; Procedure: Surgical Interventions; Procedure: non-EUS-based endoscopic procedures

INTERVENTIONS:
Procedure: Therapeutic EUS — 1. EUS-guided collection drainage (transgastric or transduodenal, performed by Lumen Apposing Metal Stents or double pigtail stents) and eventual endoscopic necrosectomy
  2. EUS-guided biliary drainage (either of the extrahepatic or intrahepatic biliary tree / transduodenal or transgastric / either as access for subsequent rendez-vous or transpapillary stenting OR for transparietal stenting by metal or plastic stents).
  3. EUS-guided gallbladder drainage via Lumen Apposing Metal Stents and eventual subsequent EUS-based cholecystolithotomy
  4. EUS-guided gastro-jejunostomy through Lumen Apposing Metal Stents
  5. EUS-directed ERCP in post-surgical anatomy (by gastro-gastrostomy or entero-enterostomy performed through Lumen Apposing Metal Stents)
  6. EUS-guided pancreatic duct drainage
  Groups: Therapeutic EUS
Procedure: Percutaneous Procedures — Procedures involving a percutaneous access to a target region (fluid collection, gallbladder, biliary tree)
  Groups: Controls
Procedure: Surgical Interventions — Surgical interventions to obtain a drainage (e.g. surgical necrosectomy, pancreatico-gastrostomy) or the bypass of a stricture (hepatico-jejunostomy or gastro-jejunostomy)
  Groups: Controls
Procedure: non-EUS-based endoscopic procedures — Other endoscopic procedures not involving EUS (enteral stenting, Enteroscopy-assisted ERCP)
  Groups: Controls

SUMMARY:
This registry aims to analyze long-term outcomes of therapeutic EUS (T-EUS) procedures, as well as to describe clinical and technical variables potentially predicting clinical success or adverse events, for a better selection of ideal candidates.

DETAILED DESCRIPTION:
This is an observational, prospective, single centre study. This registry aims to evaluate long-term clinical success of EUS-guided therapeutic interventions (T-EUS), as well as adverse events, and clinical and technical variables asociated with clinical success and adverse events.

For the purpose of this registry, the following procedures will be considered to be T-EUS procedures:

* EUS-guided collection drainage
* EUS-guided biliary drainage
* EUS-guided gallbladder drainage
* EUS-guided gastro-enterostomy
* EUS-directed ERCP
* EUS-guided pancreatic duct drainage

Each patient will be assigned to a procedure following standard clinical practice, in most instances following a routinely multidisciplinary discussion.

All patients eligible for the abovementioned clinical indications, but finally undergoing alternative procedures (e.g. surgical interventions, percutaneous interventions or other endoscopic procedures) will be proposed to be enrolled in the registry as "controls". The same variables will be collected, with the exception of technical variables related to the EUS-guided intervention.

ELIGIBILITY:
Inclusion Criteria:

* subjects candidate to therapeutic EUS (T-EUS) procedures for any underlying disease
* 18 years old or older
* able to provide an informed consent to inclusion.

Exclusion Criteria:

* age < 18 years
* inability or unwillingness to sign the informed consent form (ICF)
* contra-indication for endoscopy or use of fluoroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred for any condition treatable by therapeutic EUS procedures, benign or malignant, as first intention or after failure of other procedures.
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 30 days
  * EUS-guided collection drainage: Resolution or reduction of > 50% of fluid collections
  * EUS-guided biliary drainage: Reduction of >25% of bilirubin OR management of choledocholithiasis OR resolution of cholangitis
  * EUS-guided gallbladder drainage: Improvement of clinical symptoms or relief of inflammatory signs/symptoms related to cholecystitis
  * EUS-guided gastro-jejunostomy: Resumption of oral intake (Gastric Outlet Obstruction Scoring System >/= 2 id est at least semisolid food)
  * EUS-directed ERCP: Possibility to perform ERCP
  * EUS-guided pancreatic duct drainage: Relief of abdominal pain and reduction of analgesic drug requirement during follow-up OR reduction in the rate of recurrent pancreatitis.

SECONDARY OUTCOMES:
Adverse events | 12 months
  Any post-procedural complaint or complication requiring medical consultation or additional procedures, stratified according to American Society of Gastrointestinal Endoscopy Lexicon

OTHER OUTCOMES:
Technical success | 1 day
  Completion of the procedure through the correct positioning of the intended device in the target organ
Recurrence | 12 months
  A new onset or a worsening of the condition which was palliated through the procedure, after an initial clinical success

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Giorgio Arcidiacono, MD, FASGE, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Background] DeWitt JM, Arain M, Chang KJ, Sharaiha R, Komanduri S, Muthusamy VR, Hwang JH; AGA Center for GI Innovation and Technology. Interventional Endoscopic Ultrasound: Current Status and Future Directions. Clin Gastroenterol Hepatol. 2021 Jan;19(1):24-40. doi: 10.1016/j.cgh.2020.09.029. Epub 2020 Sep 18. PMID 32950747
- [Background] Teoh AYB, Dhir V, Kida M, Yasuda I, Jin ZD, Seo DW, Almadi M, Ang TL, Hara K, Hilmi I, Itoi T, Lakhtakia S, Matsuda K, Pausawasdi N, Puri R, Tang RS, Wang HP, Yang AM, Hawes R, Varadarajulu S, Yasuda K, Ho LKY. Consensus guidelines on the optimal management in interventional EUS procedures: results from the Asian EUS group RAND/UCLA expert panel. Gut. 2018 Jul;67(7):1209-1228. doi: 10.1136/gutjnl-2017-314341. Epub 2018 Feb 20. PMID 29463614
- [Derived] Vanella G, Frigo F, Leone R, Rossi G, Zaccari P, Stasio RC, Archibugi L, Petrone MC, Tacelli M, Palumbo D, Guazzarotti G, Bronswijk M, van Wanrooij RLJ, Guarneri G, Tamburrino D, Preatoni P, Ratti F, Catena M, Van der Merwe S, Falconi M, Capurso G, De Cobelli F, Arcidiacono PG. EUS-guided drainage of Post-Surgical versus Post-Pancreatitis collections (the RESPELL study): A prospective comparison of clinical presentations and therapeutic outcomes. Dig Liver Dis. 2026 Jan 22:S1590-8658(26)00009-5. doi: 10.1016/j.dld.2026.01.010. Online ahead of print. PMID 41577578
- [Derived] Vanella G, Frigo F, Perelli F, Bara R, Leone R, Stasio RC, Maisonneuve P, Partelli S, Aleotti F, Orsi G, Macchini M, Balzano G, Reni M, Falconi M, Capurso G, Arcidiacono PG. Long-term Outcomes of EUS-guided Gastroenterostomy (LONG-RANGE study): a prospective cohort study tracking symptom recurrence, reintervention timelines and stent modifications over time. Gastrointest Endosc. 2026 Jan 16:S0016-5107(26)00034-9. doi: 10.1016/j.gie.2026.01.007. Online ahead of print. PMID 41548724
- [Derived] Vanella G, Leone R, Frigo F, Bronswijk M, van Wanrooij RLJ, Tamburrino D, Orsi G, Belfiori G, Macchini M, Reni M, Aldrighetti L, Falconi M, Capurso G, van der Merwe S, Arcidiacono PG. Endoscopic ultrasound-guided choledochoduodenostomy versus hepaticogastrostomy combined with gastroenterostomy in malignant double obstruction (CABRIOLET_Pro): A prospective comparative study. DEN Open. 2024 Oct 6;5(1):e70024. doi: 10.1002/deo2.70024. eCollection 2025 Apr. PMID 39377069